CLINICAL TRIAL: NCT06644742
Title: The Natural History of Arrhythmogenic Cardiomyopathy With Pathogenic Plakophilin-2 Variants (PKP2-ACM): An Observational Cohort Study
Brief Title: PKP2-ACM Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-NI-A601-0124
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Genetic Diseases
Keywords: Arrhythmogenic Cardiomyopathy; Plakophilin-2; Arrhythmogenic Cardiomyopathy (AC, ARVD/C); PKP2
MeSH Terms: conditions — Cardiomyopathies; Heart Diseases; Cardiovascular Diseases; Genetic Diseases, Inborn; Arrhythmogenic Right Ventricular Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort

SUMMARY:
The goal of this study is to describe the natural history and clinical events for patients who have Arrhythmogenic Cardiomyopathy with Pathogenic Plakophilin-2 Variants (PKP2-ACM) managed with standard of care.

DETAILED DESCRIPTION:
This is an observational study with both retrospective and prospective data collection. The study is designed to describe the natural history of PKP2-ACM including the signs and symptoms, key clinical events, and impact of the disease on quality of life. A hybrid (retrospective and prospective data collection) approach is being taken with the aim of achieving robust and longitudinal data generation.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following criteria (and none of the exclusion criteria) to be eligible for study participation:

1. Male or female age 12 years or older at the time of providing informed consent (i.e., ICF provision).
2. Capable and willing to provide signed informed consent and/or assent, which includes compliance with the requirements and restrictions listed in the ICF and protocol.
3. Clinical diagnosis of arrhythmogenic cardio myopathy (ACM) as defined by the 2010 revised Task Force Criteria (TFC)
4. Documentation of a pathogenic or likely pathogenic variant in PKP2 by a CLIA-certified genetic testing laboratory
5. History of ICD implantation ≥6 months prior to ICF provision
6. Left ventricular ejection fraction by echocardiogram or cardiac magnetic resonance (CMR) ≥50% at ≤12 months prior to ICF provision

Exclusion Criteria

Patients meeting any of the following criteria are excluded from study participation:

1. Gene testing indicates that the subject's arrhythmia or cardiomyopathy may be related to a genetic etiology other than PKP2 truncating variant.
2. Concurrent participation in any other clinical investigation involving use of an investigational agent that could confound results of this study.
3. Previous participation in a study of gene transfer or gene editing.
4. NYHA Class IV heart failure.
5. Presence or requirement for mechanical circulatory support (MCS) or predicted need for MCS or heart transplantation within 6 months of enrollment.
6. Prior cardiac or other organ (lung, liver, other) transplantation.
7. Pacemaker dependent rhythm documented, as assessed by the principal investigator ≤12 months prior to enrollment.
8. Positive human immunodeficiency virus (HIV) antibody test.
9. Unwillingness to comply with study procedures, including follow-up as specified by this protocol, or unwillingness to fully cooperate with the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 12 years of age and over with confirmed PKP2-ACM.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Heart rhythm and rate monitoring measures | 36 months
  Evaluate electrophysiology as assessed by heart rate and rhythm
Cardiac biomarkers | 36 months
  Evaluate heart health as assessed by cardiac biomarkers

SECONDARY OUTCOMES:
Characterize cardiovascular events | 36 months
  Evaluate cardiovascular health as assessed by the occurrence of clinical outcomes related to the cardiovascular system
Evaluate patient reported outcomes and quality of life measures | 36 months
  Evaluate patient reported outcomes and quality of life measures through questionnaires.
Interrogate ICDs | 36 months
  Evaluate heart health as assessed by interrogation of implanted cardioverter defibrillator
Evaluate changes in health status | 36 months
  Evaluate changes in health status as assessed by occurrence of clinical outcomes
Cardiac Structure and Performance | 36 months
  Evaluating heart changes through measures of cardiac structure and performance with echocardiogram.
Evaluate genetics | Cross sectional
  Assess association with cardiomyopathy as assessed by genetic testing.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No